CLINICAL TRIAL: NCT00323895
Title: A Prospective, Randomized, Multi-Center Comparison of the CYPHER Select™ Sirolimus-Eluting Stent and Balloon Re-Angioplasty for Treatment of Patients With Intra-Des Restenosis
Brief Title: The Intra-Drug Eluting Stent (DES) Restenosis Study
Acronym: CRISTAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll - WW Leader Cardiology Clinical Research, Cordis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC05-02
Record Dates: First submitted 2006-05-09; First posted 2006-05-10 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents; Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): group with intra-Cypher™ restenosis
  Interventions: Device: drug-eluting stent and balloon angioplasty
- 2 (Active Comparator): group with intra-Taxus™ restenosis
  Interventions: Device: drug-eluting stent and balloon angioplasty
- 3 (Active Comparator): group with intra-BMS restenosis
  Interventions: Device: drug-eluting stent

INTERVENTIONS:
Device: drug-eluting stent and balloon angioplasty — CYPHER Select ™ Sirolimus-eluting Stent and any balloon brand
  Arms: 1
Device: drug-eluting stent and balloon angioplasty — CYPHER Select ™ Sirolimus-eluting Stent and any balloon brand
  Arms: 2
Device: drug-eluting stent — CYPHER Select ™ Sirolimus-eluting Stent
  Arms: 3

SUMMARY:
A Prospective, Randomized, Multi-Center Comparison of the Cypher Select™ Sirolimus-Eluting Stent and Balloon Re-Angioplasty for Treatment of Patients with Intra-Des Restenosis.

DETAILED DESCRIPTION:
This is a prospective, randomized study to be conducted at up to 33 sites in France with 3 groups of patients (1 group with intra-Taxus™ restenosis, 1 group with intra-Cypher™ restenosis and 1 control group with intra-BMS restenosis). All patients will have a repeat angiography at 9 to 12 months post-procedure and will be followed up to 12 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II-III) OR patients with documented silent ischemia;
* Patient has an intra-DES (TAXUS™ OR CYPHER™) or intra-BMS restenosis of >= 50% and <100% (by QCA online of the MLD compared to the distal reference diameter) in a native coronary artery;
* Study target lesion must be located in a restenotic native coronary artery >=2.25mm and <=3.5mm in lumen diameter and <=30mm in length by visual estimate and within a region up to 5mm to the proximal/distal stent edge;
* Study target lesion must have undergone coronary interventional treatment >= 4 weeks previously. Patients with one ore more prior PTCA procedures at the target lesion are acceptable candidates.
* Study target lesion can not be located in a vessel containing another lesion requiring treatment. Lesions located in other vessels may be treated with percutaneous revascularization at the time of the procedure, BUT they must be successfully treated prior to the treatment of the study target lesion;
* Patient is candidate for a current percutaneous revascularisation technique;
* Patient is willing to comply with the specified follow-up evaluations (including angiographic follow-up);
* Patient must provide written informed consent prior to the procedure using a form that is approved by the local Ethics Committee;

Exclusion Criteria:

* Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK >2 times normal within the preceding 72 hours and the CK enzymes remain above normal at the time of treatment;
* Has unstable angina classified as Braunwald A I-II-III;
* Unprotected left main coronary disease with ³50% stenosis;
* Significant (>50%) stenoses of additional lesions proximal or distal to the target lesion(s) that might require revascularization or impede runoff;
* Target lesion is in an internal mammary artery, saphenous vein bypass graft or is located in the left main or is ostial;
* Stent implantation(s) is a non-elective, emergency procedure;
* Stent at the target restenosed lesion is neither TAXUS™ , CYPHER™ DES nor a BMS;
* Documented left ventricular ejection fraction <=25%;
* Totally occluded vessel (TIMI 0 level).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2006-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
In stent late loss. | between 9 - 12 months

SECONDARY OUTCOMES:
In-stent, in-segment, and in-lesion binary restenosis rate by QCA. | between 9 - 12 months
In-lesion late loss as assessed by QCA. | between 9 - 12 months
In-stent and in-lesion MLD, and percent diameter stenosis (%DS) as assessed by QCA. | between 9 - 12 months
Target lesion revascularization (TLR). | 30 days, 6 and 12 months
Target vessel revascularization (TVR). | 30 days, 6 and 12 months
Target vessel failure (TVF) defined as cardiac death, myocardial infarction, or target vessel revascularization. | 30 days, 6 and 12 months
Composite of Major Adverse Cardiac Events (MACE) defined as cardiac death, myocardial infarction (Q wave and non-Q wave), emergent bypass surgery, or repeat target lesion revascularization. | 30 days, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Chevalier, MD, Principal Investigator — Centre Cardiologique du Nord, Saint Denis, France; Jean Fajadet, MD, PhD, Principal Investigator — Unité de Cardiologie Interventionnelle, Toulouse Cedex 3, France
Locations (2):
- France (2):
  - Centre Cardiologique du Nord, Saint-Denis
  - Unite de Cardiologie Interventionelle, Toulouse

REFERENCES:
- [Derived] Chevalier B, Moulichon R, Teiger E, Brunel P, Metzger JP, Pansieri M, Carrie D, Stoll HP, Wittebols K, Spaulding C, Fajadet J; Cristal Investigators. One-year results of the CRISTAL Trial, a randomized comparison of cypher sirolimus-eluting coronary stents versus balloon angioplasty for restenosis of drug-eluting stents. J Interv Cardiol. 2012 Dec;25(6):586-95. doi: 10.1111/j.1540-8183.2012.00769.x. Epub 2012 Sep 20. PMID 22994863